CLINICAL TRIAL: NCT03559543
Title: Evaluation of the Effect of the Ocoxin®-Viusid® Nutritional Supplement on the Quality of Life of Patients With Metastatic Colorectal Adenocarcinoma. Phase II
Brief Title: Evaluation of Ocoxin®-Viusid® in Metastatic Colorectal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OOS-CANCER-9
Record Dates: First submitted 2018-06-06; First posted 2018-06-18 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasm; Rectal Diseases; Colonic Diseases; Intestinal Disease; Gastrointestinal Disease; Digestive System Disease
Keywords: Nutritional supplement; Metastatic colorectal Cancer; Oxidative Stress; Ocoxin Viusid; Antioxidant
MeSH Terms: conditions — Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Rectal Diseases; Colonic Diseases; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases | interventions — Ocoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ocoxin-Viusid® (Experimental)
  Interventions: Dietary Supplement: Ocoxin-Viusid

INTERVENTIONS:
Dietary Supplement: Ocoxin-Viusid — An oral solution of Oncoxin® (30 ml vials) will be used at a rate of 60 ml daily (1 vial every 12 hours), preferably administered after breakfast and lunch. It will be prescribed for a period of 2 weeks before starting the QT up to 3 weeks after finishing the treatment.
  The treatment with Oncoxin®-Viusid® will continue in the possible periods of time of suspension of the chemotherapy treatment due to toxicities attributable to the oncospecific treatment.
  The treatment will be administered continuously for approximately 29 weeks from the patient's inclusion in the study.

SUMMARY:
The research product, registered as a nutritional supplement (Ocoxin®, oral solution), manufactured by Laboratorios Catalysis S. L., comes in the form of single-dose vials of 30 ml. It will be used at a rate of 60 ml daily (1 vial every 12 hours). Our main objective is To evaluate the effect of Ocoxin®-Viusid® on the quality of life of patients with metastatic colorectal adenocarcinoma. Our hypothesis is that the administration of the nutritional supplement Ocoxin®-Viusid® it is expected to improve the quality of life and enhance tolerance to chemotherapy in at least 70% of patients.

DETAILED DESCRIPTION:
* To evaluate the effect of Ocoxin®-Viusid® on the quality of life of patients.
* To evaluate the influence of Ocoxin®-Viusid® on tolerance to onco-specific therapy.
* Identify the changes that occur in the nutritional status of patients receiving the supplement.
* To evaluate the toxicity of Ocoxin®-Viusid® in combination with chemotherapy in patients with metastatic colorectal adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any sex, resident in Cuba, with an age greater than or equal to 18 years.
* Patients that meet the diagnostic criteria.
* Patients with general health according to Karnofsky ≥70%.
* Life expectancy greater than or equal to 3 months.
* Patients eligible to receive FOLFOX-IV chemotherapy.
* Patients who have signed the informed consent.
* Patients who have laboratory values in parameters that do not contraindicate the administration of chemotherapy:
* Hemoglobin ≥ 90 g / l
* Total Leukocyte Count ≥ 3.0 x 109 / L
* Absolute Neutrophil Count ≥1.5 x 109 / L
* Platelet Count ≥100 x 109 / L
* Total bilirubin values ≤ 1.5 times the upper limit of the normal range established in the institution.
* TGO and TGP values ≤2.5 times the upper limit of the normal interval established in the institution.
* Creatinine values within the normal limits of the institution.

Exclusion Criteria:

* Pregnant or lactating patients.
* Patients with known hypersensitivity to (5 Fluoracil, Folinic Acid or Oxaliplatin).
* Patients who are receiving another product under investigation.
* Patients with decompensated intercurrent diseases, including: hypertension, diabetes mellitus, ischemic heart disease, active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, liver damage or any other special condition that at the discretion of the doctor puts their health at risk and his life during the study or his participation in the trial.
* Patients with brain metastases.
* Patients with mental disorders that may limit adherence to the requirements of the clinical trial and may hinder the collection of information, treatment or follow-up.

It is planned to include a total of 40 patients in the study, taking into account 10% of losses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Quality of life | 8 months
  Evaluated through the European Organisation for Research and Treatment of Cancer (EORTC) CV instruments: EORTC QLQ-C30 (general quality of life in cancer patients: Physical, Role, Emotional, Cognitive, Social, Overall quality of life, Fatigue, Nausea and vomiting, Pain valorated from 1 to 4)
Quality of life | 8 months
  Evaluated through the European Organisation for Research and Treatment of Cancer (EORTC) CV instruments: QLQ-CR29 specific questionnaire of quality of life in colon cancer (Urinary frequency, Blood and mucus in stool, Stool frequency and Body image, Urinary incontinence, Dysuria, Abdominal pain, Buttock pain , Bloating, Dry mouth, Hair loss, Taste, Anxiety, Weight, Flatulence, Faecal incontinence, Sore skin, Embarrassment, Stoma care problems, Sexual interest, Impotence, Dyspareunia valorated from 1 to 4).
Tolerance of Chemotherapy | 8 months
  Treatment with chemotherapy (CT) FOLFOX-IV will be considered
Nutritional status | 8 months
  Variations in the patient's nutritional status and weight at the end of treatment will be considered

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Oncology and Radiobiology (INOR), Havana, Cuba

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Gomez EV, Perez YM, Sanchez HV, Forment GR, Soler EA, Bertot LC, Garcia AY, del Rosario Abreu Vazquez M, Fabian LG. Antioxidant and immunomodulatory effects of Viusid in patients with chronic hepatitis C. World J Gastroenterol. 2010 Jun 7;16(21):2638-47. doi: 10.3748/wjg.v16.i21.2638. PMID 20518086
- [Background] Vilar Gomez E, Sanchez Rodriguez Y, Torres Gonzalez A, Calzadilla Bertot L, Arus Soler E, Martinez Perez Y, Yasells Garcia A, Abreu Vazquez Mdel R. Viusid, a nutritional supplement, increases survival and reduces disease progression in HCV-related decompensated cirrhosis: a randomised and controlled trial. BMJ Open. 2011 Jan 1;1(2):e000140. doi: 10.1136/bmjopen-2011-000140. PMID 22021873
- [Background] Roomi MW, Roomi N, Ivanov V, Kalinovsky T, Niedzwiecki A, Rath M. Inhibition of pulmonary metastasis of melanoma b16fo cells in C57BL/6 mice by a nutrient mixture consisting of ascorbic Acid, lysine, proline, arginine, and green tea extract. Exp Lung Res. 2006 Nov-Dec;32(10):517-30. doi: 10.1080/01902140601098552. PMID 17169857
- [Background] Hernandez-Unzueta I, Benedicto A, Olaso E, Sanz E, Viera C, Arteta B, Marquez J. Ocoxin oral solution(R) as a complement to irinotecan chemotherapy in the metastatic progression of colorectal cancer to the liver. Oncol Lett. 2017 Jun;13(6):4002-4012. doi: 10.3892/ol.2017.6016. Epub 2017 Apr 10. PMID 28599406
- [Background] Maruyama T, Murata S, Nakayama K, Sano N, Ogawa K, Nowatari T, Tamura T, Nozaki R, Fukunaga K, Ohkohchi N. (-)-Epigallocatechin-3-gallate suppresses liver metastasis of human colorectal cancer. Oncol Rep. 2014 Feb;31(2):625-33. doi: 10.3892/or.2013.2925. Epub 2013 Dec 13. PMID 24337301
- [Background] Yang C, Du W, Yang D. Inhibition of green tea polyphenol EGCG((-)-epigallocatechin-3-gallate) on the proliferation of gastric cancer cells by suppressing canonical wnt/beta-catenin signalling pathway. Int J Food Sci Nutr. 2016 Nov;67(7):818-27. doi: 10.1080/09637486.2016.1198892. Epub 2016 Jun 24. PMID 27338284
- [Background] Milligan SA, Burke P, Coleman DT, Bigelow RL, Steffan JJ, Carroll JL, Williams BJ, Cardelli JA. The green tea polyphenol EGCG potentiates the antiproliferative activity of c-Met and epidermal growth factor receptor inhibitors in non-small cell lung cancer cells. Clin Cancer Res. 2009 Aug 1;15(15):4885-94. doi: 10.1158/1078-0432.CCR-09-0109. Epub 2009 Jul 28. PMID 19638461
- [Background] Siddiqui IA, Asim M, Hafeez BB, Adhami VM, Tarapore RS, Mukhtar H. Green tea polyphenol EGCG blunts androgen receptor function in prostate cancer. FASEB J. 2011 Apr;25(4):1198-207. doi: 10.1096/fj.10-167924. Epub 2010 Dec 21. PMID 21177307
- [Background] Diaz-Rodriguez E, Hernandez-Garcia S, Sanz E, Pandiella A. Antitumoral effect of Ocoxin on acute myeloid leukemia. Oncotarget. 2016 Feb 2;7(5):6231-42. doi: 10.18632/oncotarget.6862. PMID 26756220
- [Background] Hernandez-Garcia S, Gonzalez V, Sanz E, Pandiella A. Effect of Oncoxin Oral Solution in HER2-Overexpressing Breast Cancer. Nutr Cancer. 2015;67(7):1159-69. doi: 10.1080/01635581.2015.1068819. Epub 2015 Aug 4. PMID 26241555
- [Background] Bardia A, Tleyjeh IM, Cerhan JR, Sood AK, Limburg PJ, Erwin PJ, Montori VM. Efficacy of antioxidant supplementation in reducing primary cancer incidence and mortality: systematic review and meta-analysis. Mayo Clin Proc. 2008 Jan;83(1):23-34. doi: 10.4065/83.1.23. PMID 18173999
- [Background] Rodrigues MJ, Bouyon A, Alexandre J. [Role of antioxidant complements and supplements in oncology in addition to an equilibrate regimen: a systematic review]. Bull Cancer. 2009 Jun;96(6):677-84. doi: 10.1684/bdc.2009.0886. French. PMID 19493854
- [Background] Prasad KN, Hernandez C, Edwards-Prasad J, Nelson J, Borus T, Robinson WA. Modification of the effect of tamoxifen, cis-platin, DTIC, and interferon-alpha 2b on human melanoma cells in culture by a mixture of vitamins. Nutr Cancer. 1994;22(3):233-45. doi: 10.1080/01635589409514349. PMID 7877893
- [Background] Block KI, Koch AC, Mead MN, Tothy PK, Newman RA, Gyllenhaal C. Impact of antioxidant supplementation on chemotherapeutic toxicity: a systematic review of the evidence from randomized controlled trials. Int J Cancer. 2008 Sep 15;123(6):1227-39. doi: 10.1002/ijc.23754. PMID 18623084